CLINICAL TRIAL: NCT06547190
Title: Study on Treating by Eating: Role of AGEs on Mucosal Barrier and Microbiome.
Acronym: STEAMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Vlaams Instituut voor Biotechnologie (VIB) (Unknown)
Responsible Party: Principal Investigator, JoaoSabino, Prof. dr. João Sabino, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: S65600
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Advanced Glycation End products; Cooking Methods; Culinary Techniques

STUDY DESIGN:
Intervention Model Description: Randomized Cross-over Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HL (Experimental): High-to-Low AGEs diet
  Interventions: Behavioral: High AGEs diet; Behavioral: Low AGEs diet
- LH (Experimental): Low-to-High AGEs diet
  Interventions: Behavioral: High AGEs diet; Behavioral: Low AGEs diet

INTERVENTIONS:
Behavioral: High AGEs diet — Participants sequentially consumed a diet that was high in AGEs and low in AGEs just be altering their cooking method. The High AGEs diet was cooked for example by baking and grilling.
Behavioral: Low AGEs diet — Participants sequentially consumed a diet that was high in AGEs and low in AGEs just be altering their cooking method. The low AGEs diet was cooked for example by steaming and boiling.

SUMMARY:
This is an exploratory study aimed at healthy volunteers to investigate the impact of differential cooking methods on global and gut inflammation, intestinal permeability, and the gut microbiota. The investigators hypothesize that a short dietary intervention of baking and grilling of food for 2 weeks as opposed to steaming and boiling of food for 2 weeks will result in measurable differences in blood, stool and urine samples that guide towards gut and overall health and disease. All food will be provided, together with detailed cooking instructions. Food logs including photographs will be used to check whether participants complied with the study.

The investigators aim to better understand the role of cooking methods in human health, so that this can be implemented in preventive strategies and dietary treatments for specific patient groups.

DETAILED DESCRIPTION:
This is a pilot project aimed at healthy volunteers to investigate the impact of differential cooking methods on systemic and intestinal inflammation, permeability, and the gut microbiota, using a randomised cross-over design. The investigators hypothesize that a short dietary intervention of baking and grilling of food for 2 weeks (high-Advanced Glycation End Products (AGEs) diet) as opposed to steaming and boiling of food for 2 weeks (low-AGEs diet) will result in measurable differences in inflammatory, cardiometabolic and microbial markers in blood and stool as well as changes in intestinal permeability through their effect on dietary AGEs. All food will be provided, together with detailed cooking instructions. Food logs including photographs will be used to assess and check adherence to the intervention.

The investigators aim to better understand the role of cooking methods and thermal treatments in human health, so that this can be implemented in preventive strategies and dietary treatments for specific patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy
* Adhering to an omnivorous diet
* Body Mass Index (BMI) between 18.5 - 30 kg/m2
* Able to provide consent.

Exclusion Criteria:

* Participants with chronic illnesses including diabetes mellitus, cardiovascular disease, or cancer; eating disorders, irritable bowel syndrome; inflammatory bowel diseases, and previous bowel surgery (except for appendectomy).
* Current smoking
* Participants taking nonsteroidal anti-inflammatory drugs (NSAIDS), proton pump inhibitors, antacids, or laxatives one month before enrollment or antibiotics, prebiotics or probiotics six months before the start of the trial.
* Pregnancy of lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Intestinal inflammation | 2 weeks
  Measurement of faecal calprotectin through stool samples (in mg/kg)
Gut microbial metabolism | 2 weeks
  Measurement of short chain fatty acids including acetic acid, propionic acid and butyric acid through stool samples (in mg/100g stool)
Gut microbial composition | 2 weeks
  Measurement of the composition of the gut microbiota using 16s rRNA sequencing of stool samples.
Intestinal transcellular permeability | 2 weeks
  Measurement of transcellular intestinal permeability using lipopolysaccharide binding protein in blood samples
Intestinal paracellular permeability | 2 weeks
  Measurement of paracellular intestinal permeability using the lacultulose mannitol test using urine samples
Systemic inflammation | 2 weeks
  serum inflammation through OLINK inflammatory panel (measurement of 92 proteins in blood)
Systemic inflammation | 2 weeks
  Every serum CRP in blood samples (in mg/l)
Systemic cardiometabolic health | 2 weeks
  serum cardiometabolic parameters through OLINK cardiometabolic panel (measurement of 92 proteins in blood)
Systemic lipid profile | 2 weeks
  Total, LDL- and HDL-cholesterol values in blood samples (in mg/dl)
Weight changes | 2 weeks
  weight (in kg)
Handgrip strength changes | 2 weeks
  Handgrip strength (in kg)

CONTACTS AND LOCATIONS:
Overall Officials: João Sabino, MD, Principal Investigator — Leuven University Hospitals
Locations (1):
- University Hospital of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
To be discussed upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request

REFERENCES:
- [Derived] Wellens J, Vissers E, Dumoulin A, Hoekx S, Vanderstappen J, Verbeke J, Vangoitsenhoven R, Derrien M, Verstockt B, Ferrante M, Matthys C, Raes J, Verbeke K, Vermeire S, Sabino J. Cooking methods affect advanced glycation end products and lipid profiles: A randomized cross-over study in healthy subjects. Cell Rep Med. 2025 May 20;6(5):102091. doi: 10.1016/j.xcrm.2025.102091. Epub 2025 Apr 24. PMID 40280130